CLINICAL TRIAL: NCT01953913
Title: An Open Label, Multicentre, Single Arm Trial to Assess the Safety of Afatinib for Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring EGFR Mutation(s)
Brief Title: Afatinib (BIBW 2992) in Advanced Non-Small Cell Lung Cancer Patients With EGFR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.66
Record Dates: First submitted 2013-09-25; First posted 2013-10-01 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- Afatinib (Experimental): Patient will receive afatinib once daily
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Patient will receive afatinib once daily

SUMMARY:
Primary objective of the trial is to evaluate the safety of afatinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR (Epidermal growth factor receptor) mutation(s) and have never been treated with an EGFR-TKI (tyrosine kinase inhibitor). Secondary objective is to assess the time to symptomatic progression (as judged by investigator).

ELIGIBILITY:
Inclusion criteria:

* locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC)
* presence of Epidermal Growth Factor Receptor (EGFR) mutations in tumor biopsy
* male or female patients age 18 years or older (For India only, male or female patients age >=18 years and <=75 years)
* adequate organ function, defined as all of the following:

  1. Absolute Neutrophil Count (ANC) > 1500/mm3. (ANC >1000/mm3 may be considered in special circumstances such as benign cyclical neutropenia as judged by the investigator and in discussion with the sponsor).
  2. Platelet count >75,000/mm3
  3. Serum creatinine < 1.5 times of the upper limit of normal
  4. Total Bilirubin < 1.5 times upper limit of (institutional) normal (Patients with Gilbert's syndrome total bilirubin must be <4 times institutional upper limit of normal).
  5. Aspartate Amino Transferase (AST) and Alanine Amino Transferase (ALT) < three times the upper limit of (institutional) normal (ULN) (if related to liver metastases < five times ULN). 5) Eastern Cooperative Oncology Group (ECOG) score between 0 - 2 6) written informed consent by patient or guardian prior to admission into the trial that is consistent with International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP) guidelines and local law.

Exclusion criteria:

* prior treatment with an EGFR tyrosine kinase inhibitor (TKI)
* use of anti-cancer treatment within 2 weeks prior to start of trial treatment (continued use of anti-androgens and / or gonadorelin analogues for treatment of prostate cancer permitted)
* radiotherapy within 4 weeks prior to drug administration except as follows:

  1. palliative radiation to organs other than chest may be allowed up to 2 weeks prior to drug administration, and
  2. single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* major surgery within 4 weeks from day 1 of first dose of afatinib. At least 7 days should have elapsed since minor surgical procedure including placement of an access device or fine needle aspiration and at least 14 days for diagnostic or palliative video-assisted thoracoscopic surgery (VATS).
* known hypersensitivity to afatinib or any of its excipients
* history or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of >3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to starting trial treatment.
* Women of Child-Bearing Potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use medically acceptable method of contraception during the trial entry and for at least 4 weeks after treatment has ended. Adequate methods of contraception and Women of Child-Bearing Potential. Perimenopausal women must be amenorrhoeic for at least 24 months to be considered for non-childbearing potential.
* childbearing potential (see Section 4.2.3) who:

  1. are nursing or
  2. are pregnant or
  3. are not using an acceptable method of birth control, or do not plan to continue using this method throughout the trial and/or do not agree to submit to pregnancy testing required by this protocol
* history of or co-existing condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the trial or interfere with the evaluation of safety for the trial drug
* previous or concomitant malignancies at other sites, except effectively treated nonmelanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* requiring treatment with any of the prohibited concomitant medications listed, that cannot be stopped for the duration of trial participation
* known pre-existing interstitial lung disease
* presence of poorly controlled gastrointestinal disorders that could affect the absorption of the trial drug (e.g. Crohn's disease, ulcerative colitis, malabsorption, or CTC grade =2 diarrhoea of any aetiology) based on investigator assessment.
* Known active hepatitis B infection (defined as presence of Hepatitis B (HepB) sAg and/or HepB DNA), active Hepatitis C (HEP C) infection (defined as presence of Hep C RNA) and/or known Human Immunodeficiency Virus (HIV) carrier.
* meningeal carcinomatosis
* symptomatic brain metastases (patients with brain metastases, who were previously treated, are eligible provided they have asymptomatic brain metastasis for at least 4 weeks on stable doses of medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (33):
- China (12):
  - 307 Hospital of PLA, Beijing
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Jilin Province Cancer Hospital, Changchun
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Lin Yi Tumor Hospital, Linyi
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- India (14):
  - Vikram Hospital, Bangalore
  - HCG Hospital, Bengaluru
  - P VS Hospital Pvt Ltd, Calicut
  - V S Hospital, Chennai
  - Max Super Speciality Hospital, Delhi, Delhi
  - Global Hospitals, Hyderabad
  - Basavatarakam Indo - American Cancer Hospital & Research Ins, Hyderabad
  - SEAROC Cancer Centre, Jaipur
  - B. P. Poddar Hospital & Medial Research Ltd, Kolkata,West Bengal
  - Asirvatham Multispeciality Hospital, Madurai
  - Curie Manavata Cancer Centre, Maharashtra
  - Shatabdi Superspeciality Hospital, Maharashtra
  - Prince Aly Khan Hospital, Mumbai
  - Ruby Hall Clinic, Pune
- National Cancer Centre, Singapore, Singapore
- Taiwan (4):
  - E-Da Hospital, Kaohsiung City
  - NCKUH, Tainan
  - Tri-Service General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Linkou, Taoyuan

REFERENCES:
- [Derived] Zhao J, Bai H, Wang X, Wang Y, Duan J, Chen H, Xue Z, Tian Y, Cseh A, Huang DC, Wu YL, Wang J. Biomarker subset analysis of a phase IIIb, open-label study of afatinib in EGFR tyrosine kinase inhibitor-naive patients with EGFRm+ non-small-cell lung cancer. Future Oncol. 2022 Apr;18(12):1485-1497. doi: 10.2217/fon-2021-0394. Epub 2022 Feb 4. PMID 35114807
- [Derived] Tu HY, Feng J, Shi M, Zhao J, Wang Y, Chang J, Wang J, Cheng Y, Zhu J, Tan EH, Li K, Zhang Y, Lee V, Yang CT, Su WC, Lam DC, Srinivasa BJ, Rajappa S, Ho CL, Lam KC, Hu Y, Bondarde SA, Liu X, Tian Y, Xue Z, Cseh A, Huang DC, Zhou C, Wu YL. A Phase IIIb Open-Label, Single-Arm Study of Afatinib in EGFR TKI-Naive Patients with EGFRm+ NSCLC: Final Analysis, with a Focus on Patients Enrolled at Sites in China. Target Oncol. 2022 Jan;17(1):1-13. doi: 10.1007/s11523-021-00859-6. Epub 2022 Jan 12. PMID 35020119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) mutation(s), who have never been treated with an EGFR-tyrosine kinase inhibitor (TKI) were recruited in the phase IIIb open label, multicentre, single-arm trial.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that they (all participants) met all inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Afatinib: Participants received Afatinib 40 milligram (mg)/30 mg/20 mg film-coated tablets orally with 250 milliliter (mL) of water, once daily of every 28-day treatment cycle.
Period: Overall Study
Arm/Group | Afatinib
Started | 542
Treated | 541
Completed (Not discontinued from trial medication) | 0
Not Completed | 542
Not completed — Disease Progression | 349
Not completed — Worsening of underlying cancer | 22
Not completed — Adverse Event | 20
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 32
Not completed — Other than listed | 108
Not completed — Not Treated | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): It included all patients who were dispensed trial medication and documented to take at least one dose of investigational treatment (afatinib).
Arm/Group | Afatinib
Number analyzed (Participants) | 541
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286
  Male | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 537
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 541
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with serious adverse events (SAEs).
Time Frame: From first drug administration up to 28 days after last drug administration, up to 1624 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Afatinib
Number analyzed (Participants) | 541
Percentage of participants (%) | 30.3

2. Secondary Outcome: Time to Symptomatic Progression (TTSP)
Description: Time to Symptomatic progression (TTSP) was defined as time from first administration of afatinib to date of first documented clinically significant symptomatic progression that required stopping the anti-cancer treatment according to investigator's assessment. 95% confidence intervals (CIs) for the median was calculated for TTSP using Greenwood' standard error estimate.
Time Frame: From first drug administration until date of first documented clinically significant symptomatic progression that required stopping afatinib treatment, up to 1624 days.
Population: TS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib
Number analyzed (Participants) | 541
Months | 13.99 [12.91 to 15.93]

3. Secondary Outcome: Percentage of Participants With Drug-related (Afatinib-related) Adverse Events
Description: Percentage of participants with drug-related (afatinib-related) adverse events.
Time Frame: From first drug administration up to 28 days after last drug administration, up to 1624 days.
Population: TS
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Afatinib
Number analyzed (Participants) | 541
Percentage of participants (%) | 97.6

ADVERSE EVENTS:
Time Frame: For adverse events: From first drug administration up to 28 days after last drug administration, up to 1624 days. For All-cause Mortality: From first drug administration to database lock date, up to 1771 days.
Description: TS. As per the clinical trial protocol, survival follow-up was not required and was not done routinely.
Groups:
- Afatinib: Participants received Afatinib 40 milligram (mg)/30 mg/20 mg film-coated tablets orally with 250 milliliter (mL) of water, once daily of every 28- day treatment cycle.
Arm/Group | Afatinib
All-Cause Mortality (participants affected / at risk) | 46/541
Serious Adverse Events (participants affected / at risk) | 164/541
Other Adverse Events (participants affected / at risk) | 529/541
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=541)
Anaemia (Blood and lymphatic system disorders) | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac tamponade (Cardiac disorders) | 2
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 10
Duodenal obstruction (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Proctitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Vomiting projectile (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 3
General physical health deterioration (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic lesion (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pseudomonal sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Urine output decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 5
Cerebral ischaemia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 2
Coma (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Epilepsy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Speech disorder (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Ureterolithiasis (Renal and urinary disorders) | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Superior vena cava stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=541)
Anaemia (Blood and lymphatic system disorders) | 48
Diarrhoea (Gastrointestinal disorders) | 483
Mouth ulceration (Gastrointestinal disorders) | 145
Nausea (Gastrointestinal disorders) | 43
Stomatitis (Gastrointestinal disorders) | 135
Vomiting (Gastrointestinal disorders) | 54
Asthenia (General disorders) | 38
Chest pain (General disorders) | 33
Fatigue (General disorders) | 29
Mucosal inflammation (General disorders) | 57
Pyrexia (General disorders) | 43
Paronychia (Infections and infestations) | 271
Rhinitis (Infections and infestations) | 37
Upper respiratory tract infection (Infections and infestations) | 58
Urinary tract infection (Infections and infestations) | 33
Alanine aminotransferase increased (Investigations) | 77
Aspartate aminotransferase increased (Investigations) | 67
Gamma-glutamyltransferase increased (Investigations) | 36
Weight decreased (Investigations) | 70
Decreased appetite (Metabolism and nutrition disorders) | 81
Hypocalcaemia (Metabolism and nutrition disorders) | 38
Hypokalaemia (Metabolism and nutrition disorders) | 53
Back pain (Musculoskeletal and connective tissue disorders) | 48
Dizziness (Nervous system disorders) | 38
Headache (Nervous system disorders) | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 132
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 32
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 29
Dry skin (Skin and subcutaneous tissue disorders) | 47
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 41
Pruritus (Skin and subcutaneous tissue disorders) | 52
Rash (Skin and subcutaneous tissue disorders) | 383

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT01953913/SAP_000.pdf
  • Study Protocol (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT01953913/Prot_001.pdf